CLINICAL TRIAL: NCT00688090
Title: A Phase 1/2, Open Label, Non-Randomized Dose Escalation Study to Evaluate the Safety, Tolerability, Immune Response and Clinical Response of Multiple Doses of MKC1106-MT in Subjects With Advanced Melanoma
Brief Title: Safety and Immune Response to a Multi-component Immune Based Therapy (MKC1106-MT) for Patients With Melanoma.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Mihail Obrocea/Vice President-Oncology Medical & Regulatory Affairs, MannKind
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MKC1106-MT-001
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2010-08-03 (Estimated); Status verified 2010-08

CONDITIONS: Advanced Melanoma; Stage III and IV Melanoma
Keywords: Immunotherapy, Melanoma, Cancer Vaccine
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low-Dose Peptide Cohort (Experimental)
  Interventions: Biological: Biological: MKCC1106-MT
- High-Dose Peptide Cohort (Experimental)
  Interventions: Biological: Biological: MKC1106-MT

INTERVENTIONS:
Biological: Biological: MKC1106-MT — Cancer Vaccine, Immunotherapy
  Arms: High-Dose Peptide Cohort
Biological: Biological: MKCC1106-MT — Cancer Vaccine, Immunotherapy
  Arms: Low-Dose Peptide Cohort

SUMMARY:
A dose comparison of a multi-component active immunotherapy designed to stimulate an immune reaction to specific tumor associated antigens which are highly expressed on melanomas.

DETAILED DESCRIPTION:
The multi-component active immunotherapy, MKC1106-MT, consists of 1 plasmid dose and 2 peptides doses designed to stimulate an immune reaction to two tumor associated antigens (Melan-A and tyrosinase). The plasmid component will be administered on Days 1,4, 15 and 18 of each treatment cycle followed by administration of peptides on Days 29 and 32 of the treatment cycle. All components will be administered separately into superficial inguinal lymph nodes under ultrasound guidance.

ELIGIBILITY:
Inclusion Criteria:

Confirmed diagnosis of locally advanced or metastatic melanoma (American Joint Committee on Cancer [AJCC 6th edition] stage IIIB, IIIC or IV) that is refractory to standard therapy or for which no curative standard therapy exists.

Patients enrolled in the Phase 2 portion of the trial must have measurable disease by the RECIST criteria ECOG performance status of 0 or 1 Life expectancy = 3 months 18 years of age or older at screening evaluation Positive for HLA-A2, and more precisely, express A*0201 as assessed by DNA typing Tumor material from prior biopsy / surgical resection available for analysis of expression of melanoma specific antigens Adequate bone marrow reserve as evidenced by: Absolute neutrophil count (ANC) = 1,000/?L & Platelet count = 75,000/?L Adequate renal function as evidenced by: serum creatinine = 1.5 mg/dL Adequate hepatic function as evidenced by: Serum total bilirubin = 2.0 mg/dL & SGOT/SGPT = 3 times the ULN for the reference lab (= 5 the ULN for the reference lab for subjects with known hepatic metastases) Subjects must have recovered to at least baseline or Grade 1 toxicity from the effects of any prior surgery, radiotherapy or other therapies including but not limited to chemotherapy Women of childbearing potential as well as fertile men and their partners must agree to use an effective method of contraception or to abstain from sexual intercourse during the clinical trial and for 90 days following the last dose of the investigational new drug Subjects must be able to provide informed consent for participation in the clinical trial before any protocol-specific clinical trial procedure is performed

Exclusion Criteria:

No systemic infection requiring treatment Symptomatic brain metastases and/or progression of CNS metastases within the past 4 weeks; patients with treated CNS metastases (by surgery and/or radiation), who are neurologically stable, and who are no longer taking glucocorticoids, are eligible Subjects with autoimmune disorders, including, but not limited to: systemic lupus erythematosus, rheumatoid arthritis, systemic sclerosis, Sjogren's syndrome, mixed connective tissue disease, ankylosing spondylitis, Hashimoto's thyroiditis, bullous pemphigus, sarcoidosis, Behçet's syndrome, vasculitis, familial Mediterranean fever, Wegener's granulomatosis or Goodpasture's syndrome Positive HIV, hepatitis B or hepatitis C antibody test Subjects who underwent allogeneic transplant New York Heart Association Grade III or IV congestive heart failure Medical, sociological or psychological conditions that may compromise compliance or participation in the clinical trial or interfere with the interpretation of the results Subjects who have taken drugs that negatively affect immune function such as systemic corticosteroids or other immunomodulatory drugs including, but not limited to, interferon-alpha, interferon-beta, interleukin-2, etanercept, infliximab, tacrolimus, cyclosporine, mycophenolic acid, alefacept or efalizumab, within one month preceding the screening Subjects who are lactating, pregnant, or planning to become pregnant within three months of treatment completion Subjects who have received any investigational drug within the preceding four weeks of enrollment Subjects who have affected inguinal lymph nodes (metastatic process) or lack of inguinal lymph nodes (resection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2008-06; Primary Completion 2009-12 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Is to assess the safety and tolerability of MKC1106-MT regimen | 6 weeks

SECONDARY OUTCOMES:
To assess the immune response (by tetramer and ELISPOT analysis) of MKC1106-MT when administered to subjects with advanced melanoma | 6 Weeks
To determine pMEL-TYR plasmid level in the blood by PCR analysis | 6 Weeks
To determine target antigen expression (Melan A and tyrosinase) and beta2 microglobulin expression in the tumor tissue | 6 Weeks
To document any preliminary evidence of clinical response | 6 Weeks

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UCLA Medical Center, Los Angeles, California
  - H Lee Moffitt Cancer Center University of So Florida, Tampa, Florida